CLINICAL TRIAL: NCT02643810
Title: Influence of Different Types of Exercise Training on Selected Cardiovascular Parameters in Adult Individuals With Corrected Tetralogy of Fallot
Brief Title: Exercise Training in Adults With Corrected Tetralogy of Fallot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Borut Jug, Assistant Professor, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKCLRehab0012015
Record Dates: First submitted 2015-12-20; First posted 2015-12-31 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Tetralogy of Fallot
Keywords: exercise training
MeSH Terms: conditions — Tetralogy of Fallot | interventions — Exercise

ARMS (3):
- Interval training group (Active Comparator): Patients to be randomized to the 'interval training group' will have exercise training sessions 3 times per week for a period of 12 weeks. During training, they will undergo interval exercise series composed of high-intensity intervals (80-90% of peak heart rate) and low-intensity intervals (50-70% of peak heart rate).
  Interventions: Other: Exercise training
- Continuous training group (Active Comparator): Patients to be randomized to the 'continuous training group' will have exercise training sessions 3 times per week for a period of 12 weeks. They will undergo moderate continuous exercise training at 70-75% of peak heart rate.
  Interventions: Other: Exercise training
- Usual care group (No Intervention): Patients to be randomized to the 'usual care group' will undergo standard care for 12 weeks.

INTERVENTIONS:
Other: Exercise training — Patients to be randomized to the 'interval training group' or 'continuous training group' will undergo exercise training sessions 3 times per week for a period of 12 weeks.
  Arms: Continuous training group; Interval training group

SUMMARY:
In this controlled trial, patients with tetralogy of Fallot will be randomized to either interval training, continuous training, or usual care groups.

DETAILED DESCRIPTION:
Patients after surgical correction of tetralogy of Fallot (cTF) have impaired exercise tolerance as compared to healthy age-matched individuals. In this controlled trial, patients with cTF will be randomized to either interval training, continuous training, or usual care.

The aim of the study is to compare the effect of interval vs. continuous exercise training on:

i) exercise capacity ii) vascular function iii) arrhythmogenic potential iv) parameters of inflammation, hemostasis and heart failure severity v) health-related quality of life adults with cTF

ELIGIBILITY:
Inclusion Criteria:

* congenital tetralogy of Fallot surgically corrected in childhood

Exclusion Criteria:

* contraindications for exercise training,
* uncontrolled dysrhythmias,
* uncontrolled heart failure (New York Heart Association (NYHA) stage IV),
* unstable coronary or other arterial disease,
* intellectual development disorder,
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-06; Primary Completion 2017-03-05 (Actual); Study Completion 2017-03-05 (Actual)

PRIMARY OUTCOMES:
Change of maximal oxygen uptake during exercise, measured in ml/kg/min | 3 months

SECONDARY OUTCOMES:
Change of flow-mediated dilatation of the brachial artery, measured in % | 3 months
  Flow-mediated dilation (FMD) and arterial stiffness
Change of the arterial stiffness coefficient | 3 months
Change of the value of blood N terminal-proBNP, measured in ng/l | 3 months
Change of the value of blood D-dimer, measured in microg/l | 3 months
Change of the value of blood fibrinogen, measured in g/l | 3 months
Change of from-the-questionnaire-obtained quality of life, measured in points | 3 months
Change of the ECG waves | 3 months
  Estimated with digital high-resolution ECG
Change of the heart rate variability | 3 months
  Estimated with digital high-resolution ECG
Change in the result of the 6-minute walking test, measured in metres | 3 months

OTHER OUTCOMES:
Change of the heart rate recovery | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Borut Jug, MD, Ph.D., Principal Investigator — University Medical Centre Ljubljana, Slovenia
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Background] Dulfer K, Helbing WA, Duppen N, Utens EM. Associations between exercise capacity, physical activity, and psychosocial functioning in children with congenital heart disease: a systematic review. Eur J Prev Cardiol. 2014 Oct;21(10):1200-15. doi: 10.1177/2047487313494030. Epub 2013 Jun 20. PMID 23787793
- [Background] Hirth A, Reybrouck T, Bjarnason-Wehrens B, Lawrenz W, Hoffmann A. Recommendations for participation in competitive and leisure sports in patients with congenital heart disease: a consensus document. Eur J Cardiovasc Prev Rehabil. 2006 Jun;13(3):293-9. doi: 10.1097/01.hjr.0000220574.22195.d6. PMID 16926656
- [Background] Dua JS, Cooper AR, Fox KR, Graham Stuart A. Exercise training in adults with congenital heart disease: feasibility and benefits. Int J Cardiol. 2010 Jan 21;138(2):196-205. doi: 10.1016/j.ijcard.2009.01.038. Epub 2009 Feb 13. PMID 19217676
- [Background] Duppen N, Kapusta L, de Rijke YB, Snoeren M, Kuipers IM, Koopman LP, Blank AC, Blom NA, Dulfer K, Utens EM, Hopman MT, Helbing WA. The effect of exercise training on cardiac remodelling in children and young adults with corrected tetralogy of Fallot or Fontan circulation: a randomized controlled trial. Int J Cardiol. 2015 Jan 20;179:97-104. doi: 10.1016/j.ijcard.2014.10.031. Epub 2014 Oct 22. PMID 25464424
- [Background] Duppen N, Takken T, Hopman MT, ten Harkel AD, Dulfer K, Utens EM, Helbing WA. Systematic review of the effects of physical exercise training programmes in children and young adults with congenital heart disease. Int J Cardiol. 2013 Oct 3;168(3):1779-87. doi: 10.1016/j.ijcard.2013.05.086. Epub 2013 Jun 6. PMID 23746621
- [Derived] Novakovic M, Prokselj K, Rajkovic U, Vizintin Cuderman T, Jansa Trontelj K, Fras Z, Jug B. Exercise training in adults with repaired tetralogy of Fallot: A randomized controlled pilot study of continuous versus interval training. Int J Cardiol. 2018 Mar 15;255:37-44. doi: 10.1016/j.ijcard.2017.12.105. Epub 2018 Jan 3. PMID 29338917